CLINICAL TRIAL: NCT01739543
Title: A Reduction in C-section Rates Using the Hem-Avert Perianal Stabilizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stetrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PB_002
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Complications; Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational (Experimental): Subject receives Hem-Avert Device.
  Interventions: Device: Hem-Avert
- Control (No Intervention): Subject does not receive Hem-Avert Device.

INTERVENTIONS:
Device: Hem-Avert — Application of Hem-Avert
  Other Names: Hem-Avert Perianal Stabilizer
  Arms: Investigational

SUMMARY:
A REDUCTION IN C-SECTION RATES USING THE HEM-AVERT® PERIANAL STABILIZER.

DETAILED DESCRIPTION:
This study is being conducted to evaluate an existing FDA approved device called the HEM-AVERT® Perianal Stabilizer for its efficacy in reducing Cesarean births and/or reducing the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for vaginal delivery.
* Subject is willing and able to comply with the study plan as indicated by understanding and signing the Subject Informed Consent Form.
* Subjects' pre-natal examination indicates that this is to be a single birth delivery.

Exclusion Criteria:

* Subject's scheduled for vaginal delivery with anticipated complications.
* Subject is unable to understand and sign the informed consent form.
* Subject does not deliver at study facility (hospital).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Reduce C-section Rate | 24 hours
  The primary objective (purpose) of this study is to evaluate the success rate of the HEM-AVERT® device as a method of reducing C-section rates

SECONDARY OUTCOMES:
Reduce duration of 2nd stage of labor. | 24 hours
  A secondary objective is to evaluate the success rate of the HEM-AVERT® device as a method of reducing the duration of second stage of labor

CONTACTS AND LOCATIONS:
Overall Officials: Dan Burns, M.D., Principal Investigator — Unafilliated
Locations (1):
- Niagara Falls Memorial Medical Center, Niagara Falls, New York, United States

REFERENCES:
- [Derived] Burns DA. Effectiveness of a novel device in the reduction of cesarean deliveries. ISRN Obstet Gynecol. 2013 Sep 1;2013:173278. doi: 10.1155/2013/173278. eCollection 2013. PMID 24078876